CLINICAL TRIAL: NCT03890653
Title: Impact Evaluation of the Nigeria State Health Program Investment Credit (NSHPIC)
Brief Title: Impact Evaluation of the Nigeria Result-Based Financing Project
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: P128175
Record Dates: First submitted 2017-05-08; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Maternal Care Patterns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Performance-Based Financing (Experimental): At least one primary healthcare centre per ward and one General Hospital per selected LGA (in 50% of LGAs in each of the 3 states) and one secondary hospital per State will be contracted by the State Primary Health Care Development Agency ) , to deliver specified services at an agreed price. Selection of which services to focus on is based on priorities identified by the Federal Government of Nigeria and the states in 2010-2015. Initial prices for each service were based on shadow prices of providing the service and have been adjusted based on implementation experience.
  Interventions: Behavioral: Performance-Based Financing
- Decentralized Facility Financing (Experimental): In the other half of the LGA's in each treated state, at least one facility per ward will receive Decentralized Facility Financing (DFF) or equivalent financing that is not be linked to any service delivery targets. These payments would be made on a quarterly basis.
  Interventions: Behavioral: Decentralized Facility Financing
- Control (No Intervention): This is a pure control arm with no additional interventions.

INTERVENTIONS:
Behavioral: Performance-Based Financing — Incentive-based payments
  Arms: Performance-Based Financing
Behavioral: Decentralized Facility Financing — Financing not linked to service delivery.
  Arms: Decentralized Facility Financing

SUMMARY:
The World Bank and the government of Nigeria are implementing a results-based financing (RBF) project for the states of Nasarawa, Adamawa, and Ondo. This project provides incentives for improving performance at critical levels within the Nigerian health system and aims to address some of these challenges. The primary goal of the impact evaluation of this project is to determine if providing financial incentives linked directly to performance increases the quantity and quality of maternal and child health (MCH) services.

In each of the three selected States,the project finances the following interventions:

1. Performance incentives to State Government and Local Government (LGA) agencies that are triggered by Disbursement Linked Indicators (DLIs) that reflect strengthened supervision and enhanced operational support for improving health systems performance. These performance incentives would be paid out on an annual basis.
2. In half of the LGAs in each state, one facility per ward will receive Performance-Based Financing (PBF) wherein payments are made directly to individual health facilities based on the quantity and quality of a set of pre-defined services provided by each facility. These performance incentives would be paid out on a quarterly basis.
3. In the other half of the LGAs in each state one facility per ward will receive Decentralized Facility Financing (DFF) or equivalent financing that is not be linked to any service delivery targets. These payments would be made on a quarterly basis.

The evaluation of the PBF arm, which consists of making payments to health facilities conditional on performance, but within an environment of comparable levels of overall financing, will rely on experimental assignment. The effect of the PBF intervention will be identified by comparing outcomes in the LGAs receiving PBF versus those receiving DFF in the three project states. In each of these three States, the LGAs will be randomly assigned to either the PBF package or to the DFF package.

DETAILED DESCRIPTION:
A detailed description can be found in the attached project concept note.

ELIGIBILITY:
Inclusion Criteria:

1. All health facility staff in the states of Nasarawa, Adamawa and Ondo attending to maternity patients in the study period.
2. Selected mothers recently utilizing the same facilities if consent is provided.

Exclusion Criteria:

1. None.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-08-20 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Utilization of priority maternal and child health services | Each health facility assessed over a period of two days.
  The utilization of priority MCH services, as defined by the quantitative checklist used by the project to measure and reward facility performance.

SECONDARY OUTCOMES:
Utilization of priority maternal and child health services, particularly by the poor | Each health facility assessed over a period of two days.
  The utilization of priority MCH services, as defined by the quantitative checklist used by the project to measure and reward facility performance, by poor households.
Aggregated Provider Performance through Direct Clinical Observation | Each health provider assessed over a period of one day.
  We use data on direct clinical observations of labor and delivery to construct an aggregate measure of provider performance.
Aggregate Structural and Process Quality Index | Each health facility assessed over a period of two days.
  The quantitative checklist used in the government program is replicated to a large degree in the impact evaluation survey. We construct independent observations on aggregate structural and process quality measures in the same fashion as the program has constructed and rewarded.

CONTACTS AND LOCATIONS:
Overall Officials: Eeshani Kandpal, PhD, Principal Investigator — World Bank

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanna M, Loevinsohn B, Pradhan E, Fadeyibi O, McGee K, Odutolu O, Fritsche GB, Meribole E, Vermeersch CMJ, Kandpal E. Decentralized facility financing versus performance-based payments in primary health care: a large-scale randomized controlled trial in Nigeria. BMC Med. 2021 Sep 21;19(1):224. doi: 10.1186/s12916-021-02092-4. PMID 34544415